CLINICAL TRIAL: NCT05014165
Title: Backtracking Leukemia-Typical Somatic Mutations in Cord Blood
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI20N1
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (Cord Blood collection): Accrue patients with ALL and AML who indicate having banked cord blood at birth through the COG Project:EveryChild (APEC14B1)
  Interventions: Other: Cord blood Sample Collection; Other: Case identification and recruitment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cord blood Sample Collection — Obtain banked cord blood samples from consecutive childhood leukemia patients
Other: Case identification and recruitment — Cases meeting eligibility and who have given consent through APEC14B1 for future contact for non-therapeutic studies
Other: Questionnaire Administration — The family will be given an option to complete questionnaire on paper, online, or over the telephone.

SUMMARY:
A comprehensive mechanistic and epidemiological study to obtain banked cord blood samples from consecutive childhood leukemia patients enrolled in the COG Project:EveryChild (APEC14B1) study. Will attempt to backtrack the initiating genomic alteration identified in the matched diagnostic leukemia sample and molecularly characterize pre-leukemic cells. The ultimate goal of this research is to pinpoint the cell of origin of leukemogenic alterations formed in utero, elucidating the etiology of these initiating mutations (as opposed to frank leukemia), and devising a test for circulating pre-leukemia that can be applied on a population-wide basis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Aim 1: To obtain stored cord blood and dried bloodspots of pediatric leukemia patients in Project:EveryChild.

Secondary Aim 2: To conduct preliminary backtracking and characterization of ALL- and AML-typical somatic mutations in cord blood and dried bloodspots.

OUTLINE:

Accrue patients with ALL and AML who indicate having banked cord blood at birth through the APEC14B1 intake questionnaire

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a diagnosis of acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML).
* Stored diagnostic pre-treatment samples corresponding to the patient's original diagnosis of leukemia must be available for request from either the COG Biopathology Center or a treating institution
* The patient must be enrolled on APEC14B1 with consent to future contact and indicate that cord blood was stored at birth in the APEC14B1 registry intake data.
* The patient must also have been registered with COG by a North American (limited to the U.S. and Canada) member institution.
* ≤ 25 years old at the time of original diagnosis with ALL or AML
* The patient must be able to understand written and spoken English or Spanish
* All patients must provide their consent/assent, as appropriate, and for patients under the age of majority at least one parent or legal guardian must provide consent as well
* All institutional, FDA, and NCI requirements for human studies must be met

Exclusion Criteria:

* Patients who responded that cord blood was not stored at birth are excluded. Patients without stored diagnostic, pre-treatment leukemia samples at either the COG Biopathology Center or their treating institution are excluded.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patient-specific somatic alterations found in cord blood in each molecularly-defined subtype of leukemia leukemia patients in Project:EveryChild. | up to 5 years
  Investigate less common cytogenetic subtypes for which the prenatal origins have not yet been investigated.

SECONDARY OUTCOMES:
Density of alterations, calculated as # of alterations per # of cells assayed, within each flow-sorted cell population | Up to 5 years
  Determine the prenatal origins across childhood leukemia subtypes, we will perform backtracking experiments using patient-specific ddPCR probes in matched tumor and CB samples from childhood ALL and AML patients in APEC14B1 with available stored CB. To identify the cells of origin of preleukemic alterations across childhood ALL and AML subtypes, we will perform single-cell sequencing analyses in flow-sorted CB cells from patients in which a prenatal lesion has been confirmed by backtracking.

CONTACTS AND LOCATIONS:
Overall Officials: Adam de Smith, PhD, Study Chair — University of Southern California Keck School of Medicine; Logan Spector, PhD, Study Chair — University of Minnesota Masonic Cancer Center
Locations (1):
- University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota, United States